CLINICAL TRIAL: NCT06281522
Title: The Importance of Inflammatory Markers Calculated From Preoperative and Postoperative Peripheral Blood Results in the Diagnosis and Treatment of Patients Operated for Hydatid Cyst of the Lung (Lung Echinococcus Granulosus)
Acronym: Echinococcusis
Status: Recruiting | Type: Observational
Sponsor: Abdullah Adiyaman (Other)
Responsible Party: Sponsor-Investigator, Abdullah Adiyaman, Graduate Student, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Other Study IDs: University of Health Sciences
Record Dates: First submitted 2024-01-14; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Lung Hydatid Cyst
Keywords: Lung Hydatid Cyst; neutrophils,; lymphocytes,; platelets

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Operated patients with hydatid cyst of the lung — File screening and blood test results will be evaluated
  Other Names: File screening and blood test results will be evaluated

SUMMARY:
This study aims to investigate the role of these laboratory findings in the differential diagnosis and management of pulmonary hydatid cyst (PHC) by examining the number of euzonophils, neutrophils, lymphocytes, platelets and neutrophil/lymphocyte ratio, platelet/lymphocyte ratio and systemic immune inflammatory index values in the peripheral blood of patients diagnosed with pulmonary hydatid cyst (PHC) in the preoperative period and post-operative 3rd month. Although we have extensive data on hydatid liver cysts, there is limited information in the literature on the laboratory values of patients with PHC. This study aims to provide more scientific basis for the diagnosis and management of PHC and is considered as an inexpensive, reproducible and easily calculable method to improve the accurate diagnosis and management of AKH in clinical practice.

DETAILED DESCRIPTION:
Hydatid cyst of the lung (HCC) is a health problem caused by a small species of tapeworm called Echinococcus granulosus, a parasitic infection that can occur in humans and other mammals. Hydatid cysts are cysts caused by the larvae of the parasite. They most commonly form in the liver and lungs, but can also occur in other organs. E. granulosus lives in the intestines of animals and excretes them in their feces. Humans can get the eggs of this parasite through contact or under poor hygiene conditions. The ingested eggs hatch in the stomach and intestine and the larvae enter the bloodstream, then form cysts in various organs throughout the body.

Cystic echinococcosis is a disease in which a large group of patients live in conditions of material and social poverty. The disease has a widespread distribution worldwide and the regions with high disease prevalence are Southeast Europe, the Middle East, North, Central and East Asia and South America.

ELIGIBILITY:
Inclusion Criteria:

* Between January 1, 2022 - December 1, 2023, patients with hydatid cyst of the lung who were hospitalized in the Thoracic Surgery Service

Exclusion Criteria:

* Between January 1, 2022 and December 1, 2023, other patients admitted to the Thoracic Surgery Service

Ages: 18 Years to 83 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Peripheral blood results of patients hospitalized in the thoracic surgery clinic of S.B.Ü Van Training and Research Hospital due to hydatid cyst of the lung (surgery) will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Calculation of laboratory markers | 2 monts
  euzonophil (10^9/L) , neutrophil (10^9/L), lymphocyte (10^9/L), platelet (10^3/uL) counts and neutrophil/lymphocyte ratio, platelet/lymphocyte ratio, systemic immune inflammatory index (SII = P × N/L) values calculated using these data in the peripheral blood results of patients diagnosed with pulmonary hydatid cyst (PHC) in the pre-operative period and post-operative 3rd month will be examined retrospectively.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Van Training and Research Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No